CLINICAL TRIAL: NCT02248714
Title: A 4-week, Single-center, Randomized, Open-label, Parallel Group Study to Evaluate the Efficacy of Glucerna SR Using Continuous Glucose Monitoring System(CGMS) in Chinese Drug-naïve Subjects With Type 2 Diabetes
Brief Title: The Efficacy of Glucerna SR in Chinese Drug-naïve Subjects With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Yuqian Bao, Director of the Department of Endocrinology and Metabolism, Shanghai Jiao Tong University Affiliated Sixth People's Hospital, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-32
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Results first posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucerna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study arm (Experimental): Use Glucerna SR as a meal replacement at breakfast meal in the study group, meanwhile patients receive diabetes diet management (Each subject will be individually instructed by a dedicating dietitian how to implement the daily diabetes diet before starting the study.)
  Interventions: Dietary Supplement: Glucerna SR
- Control arm (No Intervention): Patients only receive diabetes diet management according to the instruction of dedicating dietitian on how to implement the daily diabetes diet.

INTERVENTIONS:
Dietary Supplement: Glucerna SR — Glucerna SR (Abbott Laboratories, Columbus, USA) is a nutritional product with lower glycemic response.
  Arms: Study arm

SUMMARY:
The purpose of the study is to evaluate the effect of Glucerna SR treating newly-diagnosed type 2 diabetes patients (NDM) on glycemic stability, with the application of CGMS (continuous glucose monitoring system) and to further realize the safety and effect of Glucerna SR on daily and day-to-day amplitude of blood glucose fluctuation.

DETAILED DESCRIPTION:
Glucerna SR (Abbott Laboratories, Columbus, USA) is a nutritional product with lower glycemic response. About 24% of the total energy provided by Glucerna SR is due to monounsaturated fatty acids, which can help keep good metabolic state in accordance with the recommendations of the American Heart Association. The aim of the study is to evaluate the effect of Glucerna SR treating newly-diagnosed type 2 diabetes patients (NDM) on glycemic stability, with the application of CGMS (continuous glucose monitoring system) and to further realize the safety and effect of Glucerna SR consumed as a meal replacement at breakfast meal on daily and day-to-day amplitude of blood glucose fluctuation.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed type 2 diabetes mellitus
* FPG≤13mmol/l and/or 2hPG≤18mmol/l
* HbA1c≥7.0%
* BMI (Body Mass Index)≥18.5kg/m2

Exclusion Criteria:

* Patients taking any class of injectible or oral hypoglycemia agents to manage their hyperglycemia.
* Female patients are in gestation, lactation or intend to be pregnant in the study period.
* Patients are with type 1 diabetes, or other special types of diabetes, or gestational diabetes mellitus.
* Patients with drug hypersensitivity.
* Patients with obvious hepatic or renal diseases (ALT, T-Bil>1.5 times of upper limit)
* Patients with severe or unstable angina, or heart failure (NYHA class III/IV)
* Patients having acute complications, or chronic complications maintained insulin therapy or insulin therapy under stress.
* Patients with chronic consumptive diseases like cerebrovascular disease, tumor, tuberculosis, or hematopathy, psychosis, autoimmune disease or severe digestive dysfunction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2014-03; Primary Completion 2018-06 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuqian Bao, MD, Principal Investigator — Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Locations (1):
- Shanghai Jiao Tong University Affiliated Sixth People's Hospital, Shanghai, Shanghai Municipality, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Arm | Control Arm
Started | 66 | 65
Completed | 62 | 61
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Arm | Control Arm | Total
Number analyzed (Participants) | 62 | 61 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (9.1) | 56.5 (8.4) | 56.7 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 25 | 57
  Male | 30 | 36 | 66
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 24.6 (3.0) | 25.3 (2.9) | 24.9 (2.9)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 131.7 (14.8) | 128.9 (12.1) | 130.4 (13.6)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 80.4 (9.2) | 79.7 (9.0) | 80.1 (9.1)
Total Cholesterol (TC) [Mean (Standard Deviation); unit: mmol/l] | 5.1 (0.8) | 5.1 (1.0) | 5.1 (0.9)
Triglycerides [Mean (Standard Deviation); unit: mmol/l] | 1.9 (1.6) | 1.6 (0.6) | 1.7 (1.2)
High Density Lipoprotein Cholesterol(HDL-c) [Mean (Standard Deviation); unit: mmol/l] | 1.2 (0.3) | 1.2 (0.2) | 1.2 (0.3)
Low Density Lipoprotein Cholesterol(LDL-c) [Mean (Standard Deviation); unit: mmol/l] | 3.2 (0.8) | 3.2 (0.8) | 3.2 (0.8)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mmol/l] | 7.4 (0.8) | 7.4 (1.2) | 7.4 (1.0)
2-h Plasma Glucose (2h-PG) [Mean (Standard Deviation); unit: mmol/l] | 15.0 (2.7) | 15.0 (2.6) | 15.0 (2.6)
Glycated Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage of glycated hemoglobin A1c] | 7.2 (0.6) | 7.2 (0.6) | 7.2 (0.6)
Glycated Albumin (GA) [Mean (Standard Deviation); unit: percentage of glycated albumin] | 18.1 (2.8) | 17.7 (2.9) | 17.9 (2.8)
Homeostasis Model Assessments of Insulin Resistance (HOMA-IR) [Mean (Standard Deviation); unit: mU/L*mmol/L] | 4.2 (2.9) | 4.3 (2.4) | 4.3 (2.6)
Incremental AUC of Postprandial Blood Glucose (AUCpp) [Mean (Standard Deviation); unit: min*mmol/l] | 522.5 (335.9) | 479.4 (236.8) | 501.1 (290.6)
Standard Deviation of Blood Glucose (SDBG) [Mean (Standard Deviation); unit: mmol/l] | 1.9 (0.7) | 1.8 (0.6) | 1.8 (0.7)
Mean Amplitude of Glycaemic Excursions (MAGE) [Mean (Standard Deviation); unit: mmol/l] | 5.0 (2.0) | 4.8 (1.7) | 4.9 (1.9)
Glucose Coefficient of Variation(CV) [Mean (Standard Deviation); unit: percentage of CV] — glucose coefficient of variation (CV) was calculated by dividing the standard deviation of blood glucose values by the mean of the corresponding glucose readings.
  percentage of CV | 21.5 (7.3) | 20.9 (5.6) | 21.2 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in AUCpp
Description: Subjects will perform continues blood glucose monitoring using CGMS for 72 hours at the beginning of the study and within the last three days during a 4-week treatment interval and AUCpp based on CGMS data was calculated as the area between the glucose concentration-time curve, and the pre-prandial baseline glucose value measured at 4 h after each meal.
Time Frame: 4 weeks
Population: The analysis population is subjects who completed the whole study.
Measure: Mean (Standard Deviation); unit: min*mmol/L
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 62 | 61
min*mmol/L | -287.8 (368.7) | -31.2 (301.6)

2. Primary Outcome: Change From Baseline in SDBG
Description: Subjects will perform continues blood glucose monitoring using CGMS for 72 hours at the beginning of the study and within the last three days during a 4-week treatment interval and SDBG will be calculated based on CGMS data.
Time Frame: 4 weeks
Population: The analysis population is subjects who completed the whole study.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 62 | 61
mmol/L | -0.6 (0.8) | -0.2 (0.7)

3. Primary Outcome: Change From Baseline in MAGE
Description: Subjects will perform continues blood glucose monitoring using CGMS for 72 hours at the beginning of the study and within the last three days during a 4-week treatment interval and MAGE will be calculated based on CGMS data.
Time Frame: 4 weeks
Population: The analysis population is subjects who completed the whole study.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 62 | 61
mmol/L | -1.6 (2.3) | -0.6 (2.1)

4. Primary Outcome: Change From Baseline in Glucose Coefficient of Variation(CV)
Description: Subjects will perform continues blood glucose monitoring using CGMS for 72 hours at the beginning of the study and within the last three days during a 4-week treatment interval and glucose coefficient of variation(CV) will be calculated based on CGMS data dividing the standard deviation of blood glucose values by the mean of the corresponding glucose readings.
Time Frame: 4 weeks
Population: The analysis population is subjects who completed the whole study.
Measure: Mean (Standard Deviation); unit: percentage of CV
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 62 | 61
percentage of CV | -4.7 (8.1) | -0.2 (7.6)

5. Secondary Outcome: Change From Baseline in BMI
Description: the change of BMI between the end and the beginning of the study
Time Frame: 4 weeks
Population: The analysis population is subjects who completed the whole study.
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 62 | 61
kg/m2 | -0.5 (0.5) | -0.5 (0.5)

6. Secondary Outcome: Change From Baseline in Systolic Blood Pressure
Description: the change of systolic blood pressure between the end and the beginning of the study
Time Frame: 4 weeks
Population: The analysis population is subjects who completed the whole study.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 62 | 61
mmHg | -7.5 (11.8) | -2.8 (14.0)

7. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure
Description: the change of diastolic blood pressure between the end and the beginning of the study
Time Frame: 4 weeks
Population: The analysis population is subjects who completed the whole study.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 62 | 61
mmHg | -4.4 (10.8) | -1.1 (8.8)

8. Secondary Outcome: Change From Baseline in TC
Description: the change of total cholesterol between the end and the beginning of the study
Time Frame: 4 weeks
Population: The analysis population is subjects who completed the whole study.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 62 | 61
mmol/L | -0.1 (0.7) | -0.2 (0.7)

9. Secondary Outcome: Change From Baseline in Triglycerides
Description: the change of triglycerides between the end and the beginning of the study
Time Frame: 4 weeks
Population: The analysis population is subjects who completed the whole study.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 62 | 61
mmol/L | -0.4 (1.3) | -0.2 (0.5)

10. Secondary Outcome: Change From Baseline in HDL-c
Description: the change of HDL-c between the end and the beginning of the study
Time Frame: 4 weeks
Population: The analysis population is subjects who completed the whole study.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 62 | 61
mmol/L | -0.0 (0.1) | 0.0 (0.1)

11. Secondary Outcome: Change From Baseline in LDL-c
Description: the change of LDL-c between the end and the beginning of the study
Time Frame: 4 weeks
Population: The analysis population is subjects who completed the whole study.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 62 | 61
mmol/L | -0.1 (0.6) | -0.1 (0.6)

12. Secondary Outcome: Change From Baseline in FPG
Description: the change of FPG between the end and the beginning of the study
Time Frame: 4 weeks
Population: The analysis population is subjects who completed the whole study.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 62 | 61
mmol/L | -0.7 (0.9) | -0.6 (1.0)

13. Secondary Outcome: Change From Baseline in 2h-PG
Description: the change of 2h-PG between the end and the beginning of the study
Time Frame: 4 weeks
Population: The analysis population is subjects who completed the whole study.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 62 | 61
mmol/L | -2.9 (3.3) | -2.0 (3.1)

14. Secondary Outcome: Change From Baseline in HbA1c
Description: the change of HbA1c between the end and the beginning of the study
Time Frame: 4 weeks
Population: The analysis population is subjects who completed the whole study.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 62 | 61
percentage of HbA1c | -0.5 (0.4) | -0.5 (0.4)

15. Secondary Outcome: Change From Baseline in GA
Description: the change of GA between the end and the beginning of the study
Time Frame: 4 weeks
Population: The analysis population is subjects who completed the whole study.
Measure: Mean (Standard Deviation); unit: percentage of GA
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 62 | 61
percentage of GA | -2.3 (2.6) | -1.8 (2.9)

16. Secondary Outcome: Change From Baseline in HOMA-IR
Description: the change of HOMA-IR between the end and the beginning of the study
Time Frame: 4 weeks
Population: The analysis population is subjects who completed the whole study.
Measure: Mean (Standard Deviation); unit: mU/L*mmol/L
Arm/Group | Study Arm | Control Arm
Number analyzed (Participants) | 62 | 61
mU/L*mmol/L | -1.3 (2.2) | -1.0 (1.9)

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: The subjects are newly diagnosed and untreated T2D, so they are not prone to hypoglycemia.
Arm/Group | Study Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/65
Other Adverse Events (participants affected / at risk) | 0/66 | 0/65

LIMITATIONS AND CAVEATS:
1.The intervention period was relatively short. 2. The open-label design of the current study may introduce some extent of bias. 3.Only untreated T2D patients were admitted in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-31): https://cdn.clinicaltrials.gov/large-docs/14/NCT02248714/Prot_SAP_000.pdf